CLINICAL TRIAL: NCT03513575
Title: Comparison of Five Different Salivary Buffering Agents on the Changes in pH of Saliva in a Cohort Previously Exposed to a Test Sweetened Flavored Milk Drink: A Randomized Controlled Crossover Trial
Brief Title: Comparison of 5 Buffering Agents on Changes in Salivary pH in Individuals Previously Exposed to a Test Flavoured Milk
Acronym: SALPH-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Meru S (Other)
Responsible Party: Sponsor-Investigator, Dr Meru S, Prof & Head, Dept of Oral Medicine & Radiology, Uttaranchal Dental & Medical Research Institute
Organization: Uttaranchal Dental & Medical Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UDMRI_Sal_pH_M; U1111-1212-4324 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2018-04-17; First posted 2018-05-01 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Saliva Altered; Oral Hygiene; pH; Tooth Structure; Disorder
Keywords: pH of saliva; Flavored Milk; buffering agent; oral hygiene
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: only primary investigator will know the intervention done by the subject. The outcome investigator(assessor) will be unaware (blinded) to which intervention the subject is undertaken.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1: no intervention (Active Comparator): The subject collects the unstimulated saliva in a sterile glass dish for the measurement of baseline pH of the saliva. The subject is then given 100 ml of test flavored milk drink, Amul Kool® milk, (Gujarat Cooperative Milk Marketing Federation Ltd.) to drink. The subject will sip, swish and swallow the drink within 2 minutes.
  Unstimulated saliva samples are collected from the subject to measure the pH of saliva after 5, 15, 30, 45 and 60 minutes of consumption of the test flavored milk drink.
  Interventions: Other: Group 1: no intervention
- Group 2: tap water gargle (Experimental): The subject collects the unstimulated saliva in a sterile glass dish for the measurement of baseline pH of the saliva. The subject is then given 100 ml of test flavored milk drink, Amul Kool® milk, (Gujarat Cooperative Milk Marketing Federation Ltd.) to drink. The subject will sip, swish and swallow the drink within 2 minutes.
  Unstimulated saliva samples are collected from the subject to measure and record the pH of saliva after 5 and 15 minutes of consumption of the test flavored milk drink.
  The subject will use 10 ml of tap water as mouth rinse to swish for 60 seconds and spit. Unstimulated saliva samples are collected from the subject to measure and record the pH of saliva at 15, 30 and 45 minutes after the subject completes the gargle as an intervention.
  Interventions: Other: Group 2: tap water gargle
- Group 3: 0.2% chlorhexidine (Experimental): The subject collects unstimulated saliva in a sterile glass dish for measurement of baseline pH of saliva. The subject is then given 100ml of test flavored milk drink, Amul Kool® milk, (Gujarat Cooperative Milk Marketing Federation Ltd.) to drink. The subject will sip, swish and swallow the drink within 2 minutes.Unstimulated saliva samples are collected from the subject to measure and record the pH of saliva after 5 and 15 minutes of consumption of the test flavored milk drink.
  The subject will use 10 ml of 0.2% Chlorhexidine mouthrinse (Rexidine®, Indoco Remidies Ltd, Mumbai, India) to swish for 60 seconds and spit. Unstimulated saliva samples are collected thereafter to measure and record the pH of saliva at 15, 30 and 45 minutes after subject completes the gargle as an intervention.
  Interventions: Other: Group 3: 0.2% Chlorhexidine
- Group 4: fluoridated tooth paste (Experimental): The subject collects unstimulated saliva in a sterile glass dish for measurement of baseline pH of saliva. The subject is then given 100 ml of test flavored milk drink, Amul Kool® milk, (Gujarat Cooperative Milk Marketing Federation Ltd.) to drink. The subject will sip, swish and swallow the drink within 2 minutes. Unstimulated saliva samples are collected from the subject to measure and record the pH of saliva after 5 and 15 minutes of consumption of the test flavored milk drink.
  The subject will brush with fluoridated toothpaste (Colgate Total®, Colgate-Palmolive Co., Mumbai, India) for 2 minutes using soft brush. Unstimulated saliva samples are collected thereafter to measure and record the pH of saliva at 15, 30 and 45 minutes after subject completes the brushing as an intervention.
  Interventions: Other: Group 4: Fluoridated tooth paste
- Group 5: Polyol containing gum (Experimental): The subject collects unstimulated saliva in a sterile glass dish for the measurement of baseline pH of saliva. The subject is then given 100 ml of test flavored milk drink, Amul Kool® milk, (Gujarat Cooperative Milk Marketing Federation Ltd.) to drink. The subject will sip, swish and swallow the drink within 2 minutes. Unstimulated saliva samples are collected from the subject to measure and record the pH of saliva after 5 and 15 minutes of consumption of the test flavored milk drink.
  The subject will chew polyol containing gum (Orbit®, Wrigley Company) for 5 minutes and spit. Unstimulated saliva samples are thereafter collected from to measure and record the pH of saliva at 15, 30 and 45 minutes after the subject completes the chewing gum as an intervention.
  Interventions: Other: Group 5: Polyol containing gum
- Group 6: 1% sodium bicarbonate solution (Experimental): The subject collects the unstimulated saliva in a sterile glass dish for the measurement of baseline pH of the saliva. The subject is then given 100 ml of test flavored milk drink, Amul Kool® milk, (Gujarat Cooperative Milk Marketing Federation Ltd.) to drink. The subject will sip, swish and swallow the drink within 2 minutes.
  Unstimulated saliva samples are collected from the subject to measure and record the pH of saliva after 5 and 15 minutes of consumption of the test flavored milk drink.
  The subject will use 10 ml freshly prepared 1% sodium bicarbonate w/v solution to swish for 60 seconds and spit.
  Unstimulated saliva samples are collected from the subject to measure and record the pH of saliva at 15, 30 and 45 minutes after the subject completes the gargle as an intervention.
  Interventions: Other: Group 6: 1% sodium bicarbonate solution

INTERVENTIONS:
Other: Group 1: no intervention — Unstimulated saliva samples are collected from the subject to measure the pH of saliva after 5, 15, 30, 45 and 60 minutes of consumption of the test flavored milk drink without any intervention.
  Arms: Group 1: no intervention
Other: Group 2: tap water gargle — The subject will use 10 ml of tap water as mouth rinse to swish for 60 seconds and spit, 15minutes after the subject has consumed the test flavored milk drink. Unstimulated saliva samples are collected from the subject to measure and record the pH of saliva at 15, 30 and 45 minutes after the subject completes the gargle as an intervention.
  Arms: Group 2: tap water gargle
Other: Group 3: 0.2% Chlorhexidine — The subject will use 10 ml of 0.2% Chlorhexidine mouth rinse (Rexidine®, Indoco Remidies Ltd, Mumbai, India) to swish for 60 seconds and spit, 15minutes after the subject has consumed the test flavored milk drink. Unstimulated saliva samples are collected from the subject to measure and record the pH of saliva at 15, 30 and 45 minutes after the subject completes the gargle as an intervention.
  Arms: Group 3: 0.2% chlorhexidine
Other: Group 4: Fluoridated tooth paste — The subject will Brush with fluoridated toothpaste-(Colgate Total®, Colgate-Palmolive Company, Mumbai, India) for 2 minutes using soft brush, 15minutes after the subject has consumed the test flavored milk drink. Unstimulated saliva samples are collected from the subject to measure and record the pH of saliva at 15, 30 and 45 minutes after the subject completes using tooth paste as an intervention.
  Arms: Group 4: fluoridated tooth paste
Other: Group 5: Polyol containing gum — The subject will chew polyol containing gum (Orbit®, WrigleyCompany) for 5 minutes and spit, 15minutes after the subject has consumed the test flavored milk drink. Unstimulated saliva samples are collected from the subject to measure and record the pH of saliva at 15, 30 and 45 minutes after the subject completes chewing as an intervention.
  Arms: Group 5: Polyol containing gum
Other: Group 6: 1% sodium bicarbonate solution — The subject will use 10 ml freshly prepared 1% sodium bicarbonate w/v solution to swish for 60 seconds and spit, 15minutes after the subject has consumed the test flavored milk drink. Unstimulated saliva samples are collected from the subject to measure and record the pH of saliva at 15, 30 and 45 minutes after the subject completes the gargle as an intervention.
  Arms: Group 6: 1% sodium bicarbonate solution

SUMMARY:
The diurnal variation in the flow of saliva and hence the composition of saliva is an established fact. Consumption of most types of acidic and sweetened foods and beverages are known to reduce the pH of saliva and some of them even reduce it to critical pH levels and result in structural damage to the hard tissues of the tooth.

The purpose of this study is to ascertain the effect of the selected commercially available test sweetened flavored milk drink on the salivary pH and assess the buffering capacity of the saliva with or without various intervention measures following the exposure to the test flavored milk drink at different time intervals.

DETAILED DESCRIPTION:
There are substantial existing evidences that there is diurnal variation in the flow of saliva and hence the composition of saliva. The average of normal pH of saliva is reported to be 6.8. Consumption of most types of acidic and sweetened foods and beverages are known to reduce the pH of saliva and some of them even reduce it to critical pH levels and result in structural damage to the hard tissues of the tooth.

Such damages can be prevented by maintaining the pH of saliva within optimal range by using oral hygiene measures.

The purpose of this study is to ascertain the effect of the selected commercially available test sweetened flavored milk drink containing sugar on the pH of saliva and assess the buffering capacity of the saliva with or without various intervention measures following the exposure to the test flavored milk drink at different time intervals.

Aims and Objectives:

1. To measure the pH of saliva post-exposure to test sweetened flavored milk drink after 5, 15, 30, 45 and 60 minutes.
2. To measure the pH of saliva at 15, 30 and 45 minutes after using a tap water gargle as a buffering agent in those subjects who had prior exposure to test sweetened flavored milk drink 15 minutes ago.
3. To measure the pH of saliva at 15, 30 and 45 minutes after using a 0.2%Chlorhexidine mouth rinse as a buffering agent in those subjects who had prior exposure to test sweetened flavored milk drink 15 minutes ago.
4. To measure the pH of saliva at 15, 30 and 45 minutes after chewing Orbit® gum as a buffering agent in those subjects who had prior exposure to test sweetened flavored milk drink 15 minutes ago
5. To measure the pH of saliva at 15, 30 and 45 minutes after brushing with fluoridated tooth paste and soft brush as a buffering agent in those subjects who had prior exposure to test sweetened flavored milk drink 15 minutes ago
6. To measure the pH of saliva at 15, 30 and 45 minutes after gargling with 1% solution of baking soda as a buffering agent in those subjects who had prior exposure to test sweetened flavored milk drink 15 minutes ago
7. To compare the efficacy of buffering agents on the pH of saliva at 15, 30, 45 minutes post intervention in subjects who have had the test flavored milk drink 15 min prior to the a specific intervention, with the pH of saliva recorded in the same subjects at the same time periods when no intervention with any buffering agent was carried out after having the test sweetened flavored milk drink.
8. To compare the pH of saliva recorded in the subjects at 15, 30, 45 minutes time periods when they used an intervention of gargle with tap water, with that recorded when they used mouth rinse of 0.2% Chlorhexidine, with that recorded when they brushed with soft brush and fluoridated tooth paste, with that recorded when they gargled with 1% baking soda solution and with that recorded when they chewed Orbit® chewing gum (15 minutes after using the test sweetened flavored milk drink)

Materials and Methods:

30 volunteers in the age group of 18- 30 year with healthy oral cavities will be selected. Subjects with a history of any chronic medical illness, history of allergy, intake of drugs in the last 8 weeks, history of gastritis, bulimia will be excluded. Subjects with a DMFT score of more than 2 and Loe and Sillness Index of more than 0 will be excluded. Individuals who have and are currently undergoing orthodontic treatment will not be included in the study. Individuals who smoke or chew tobacco will not be included in the study sample. An informed consent for the research will be obtained from all the subjects who have volunteered for the study. The trial will be conducted as per the guidelines in the WHO-Handbook for Good Clinical Practice and the research protocol is approved by the Institutional Ethics Committee of the college.

The test flavored milk drink that will be selected is Amul Kool® (Gujarat Cooperative Milk Marketing Federation Ltd)

The various buffering agents that will be used are:

1. 0.2% Chlorhexidine mouth wash (Rexidine®, Indoco Remidies Ltd, Mumbai, India)- 10 ml solution swish for 60 sec and spit
2. Tap water- 10ml swish for 60 sec and spit
3. Brushing with fluoridated (Colgate Total®, Colgate-Palmolive Company, Mumbai, India) tooth paste- 2min using soft brush
4. Chewing polyol containing gum (Orbit®, Wrigley Company)- chew for 5 minutes and spit
5. Freshly prepared Sodium bicarbonate (baking soda) 1% w/v solution swish for 60 sec and spit.

The observer who will be recording the salivary pH will remain blinded about the samples and buffering agent used.

The select individuals will be instructed to not use any mouth wash as part of oral hygiene regimen on test day and not consume any food or beverage for 2 hours prior to the collection of baseline sample of saliva at 10 AM on the test day. The select group of 30 individuals will be given a sample of 100 ml of the test sweetened flavored milk drink after recording their baseline salivary pH (0 min). They will be asked to sip, swish and swallow the drink within 2 minutes. After the exposure, salivary samples will be collected at 5 min and 15 min intervals for assessment of pH. Fifteen minutes after the exposure (consumption of test drink), the individuals will be asked to use one of the intervention methods included in this study. The salivary samples will be collected after 15, 30 and 45 minutes interval after the intervention. (i.e. 30, 45 and 60 minutes post exposure to the test drink respectively) The same protocol will be repeated using each intervention methods included in this study after a wash out period of minimum of 3 days. The protocol will be repeated on the study sample without any intervention following the exposure to the test sweetened flavoured milk as a control.

Measurement of salivary pH will be done using a portable PH-035 Digital pH meter with automatic temperature compensation, to the accuracy of 0.1 and the machine will be calibrated on the morning of every test day and after 60 uses during the test day using Aquasol® pH calibration solutions with pH 4, 7 and 10.

ELIGIBILITY:
Inclusion Criteria:

* subjects in the age group of 18 to 30 years.
* subjects with a DMFT index score of less than 2.
* subjects with Loe and Silness index score of 0.
* subjects willing to volunteer for the study.
* subjects who are available for the whole study period of 4 months

Exclusion Criteria:

* subjects with history of gastritis and bulimia.
* subjects with chronic medical illness.
* subjects with history of allergy.
* subjects with history of drug intake for last 8 weeks.
* subjects who smoke or chew tobacco.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
pH of saliva at baseline | 0 minute
  All subjects in all groups collects the unstimulated saliva in a sterile glass dish for the measurement of baseline pH of the saliva. The subject will give the saliva sample just before being exposed to the test mixed fruit juice by swishing 100ml of Amul Kool® Flavored Milk drink in mouth for 2 minutes and then drinking it The outcome accessor is blinded to origin of sample (from which group).

SECONDARY OUTCOMES:
pH of Saliva 5 minutes after exposure to test flavored milk drink | 5 minutes
  All subjects will be given 100 ml of test flavored milk drink, Amul Kool® Milk to drink. The subject will sip, swish and swallow the drink within 2 minutes. Five minutes after this, each subject will give unstimulated saliva in a sterile dish for measurement of saliva - 5minutes after exposure to test flavored milk drink. The outcome accessor is blinded to the origin of sample (from which group).
pH of Saliva 15 minutes after exposure to test flavored milk drink | 15 minutes
  All subjects will be given 100 ml of test flavored milk drink, Amul Kool® Milk to drink. The subject will sip, swish and swallow the drink within 2 minutes. Fifteen minutes after this, each subject will give unstimulated saliva in a sterile dish for measurement of saliva - 15minutes after exposure to test flavored milk drink. The outcome accessor is blinded to the origin of sample (from which group).
pH of Saliva 30 minutes after exposure to test flavored milk drink | 30 minutes
  All subjects from all six (5 experimental and 1 comparator) groups will perform assigned intervention at time 15minutes post exposure to test flavored milk drink, Amul Kool® Milk and shall give unstimulated saliva in a sterile dish for measurement of pH -30minutes after exposure to test flavored milk drink or in other words 15minutes after assigned intervention. The outcome accessor is blinded to origin of sample (from which group).
pH of Saliva 45 minutes after exposure to test flavored milk drink | 45 minutes
  All subjects from all six (5 experimental and 1 comparator) groups will perform assigned intervention at time 15minutes post exposure to test flavored milk drink, Amul Kool® Milk and shall give unstimulated saliva in a sterile dish for measurement of pH -45minutes after exposure to test flavored milk drink or in other words 30minutes after assigned intervention. The outcome accessor is blinded to origin of sample (from which group).
pH of Saliva 60 minutes after exposure to test flavored milk drink | 60 minutes
  All subjects from all six (5 experimental and 1 comparator) groups will perform assigned intervention at time 15minutes post exposure to test flavored milk drink, Amul Kool® Milk and shall give unstimulated saliva in a sterile dish for measurement of pH -60minutes after exposure to test flavored milk drink or in other words 45minutes after assigned intervention. The outcome accessor is blinded to origin of sample (from which group).

CONTACTS AND LOCATIONS:
Overall Officials: Meru S, MDS, Principal Investigator — Uttaranchal Dental & Medical Research Institute
Locations (1):
- Department of Oral Medicine & Radiology, Uttaranchal Dental & Medical Research Institute, Dehradun, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sudeep C B, Vipin Jain, Mathew Maliyil , Peter Simon Sequeira, Jithesh Jain. Effects on pH Value of Saliva Following Intake of Three Beverages Containing Apple Juice - A Double Blind Cross- Over Study. National Journal of Medical and Dental Research 1(4): 18-23,2013
- [Background] Choi SE, Kim HS. Sodium Bicarbonate Solution versus Chlorhexidine Mouthwash in Oral Care of Acute Leukemia Patients Undergoing Induction Chemotherapy: A Randomized Controlled Trial. Asian Nurs Res (Korean Soc Nurs Sci). 2012 Jun;6(2):60-6. doi: 10.1016/j.anr.2012.05.004. Epub 2012 May 24. PMID 25030829
- [Background] Chandel S, Khan MA, Singh N, Agrawal A, Khare V. The effect of sodium bicarbonate oral rinse on salivary pH and oral microflora: A prospective cohort study. Natl J Maxillofac Surg. 2017 Jul-Dec;8(2):106-109. doi: 10.4103/njms.NJMS_36_17. PMID 29386812
- [Background] Margaret F. Lemaster. Restore pH balance. Sunstar spotlight, special sponsored supplement. March 2012
- [Background] Bhavna Jha Kukreja, Vidya Dodwad, Herbal mouth washes- a gift of nature. International Journal of Pharma and Bio Sciences 3(2);46-52:2012
- [Background] de Almeida Pdel V, Gregio AM, Machado MA, de Lima AA, Azevedo LR. Saliva composition and functions: a comprehensive review. J Contemp Dent Pract. 2008 Mar 1;9(3):72-80. PMID 18335122
- [Background] Chitharanjan Shetty, Mitra N Hegde, Darshana Devadiga.Correlation between dental caries with salivary flow, pH and buffering capacity in adult south Idoan population: An in-vitro study.Internationl J Res Ayurveda Pharm 4(2):219-223,2013
- [Background] Tenuta LM, Fernandez CE, Brandao AC, Cury JA. Titratable acidity of beverages influences salivary pH recovery. Braz Oral Res. 2015;29:S1806-83242015000100234. doi: 10.1590/1807-3107BOR-2015.vol29.0032. Epub 2015 Feb 11. PMID 25715032
- [Background] Sudeep CB, Anzil KS Ali, Vivek S, Ambalavanan P, Vivek Suku Ninan, Fajar Ummer. Effects on ph value of saliva following intake of three beverages: A double blind cross-over study. International Journal of Dental and Health Sciences.1(3);18-23:2013
- [Background] Dawes C. What is the critical pH and why does a tooth dissolve in acid? J Can Dent Assoc. 2003 Dec;69(11):722-4. PMID 14653937
- [Background] Ciolino LA, McCauley HA, Fraser DB, Wolnik KA. The relative buffering capacities of saliva and moist snuff: implications for nicotine absorption. J Anal Toxicol. 2001 Jan-Feb;25(1):15-25. doi: 10.1093/jat/25.1.15. PMID 11215994
- [Background] Larsen MJ, Nyvad B. Enamel erosion by some soft drinks and orange juices relative to their pH, buffering effect and contents of calcium phosphate. Caries Res. 1999;33(1):81-7. doi: 10.1159/000016499. PMID 9831784
- [Background] Hayden, Madison R., The Effect of Cheese on the pH Levels in the Oral Cavity. Honors College Capstone Experience/Thesis Projects. Paper 563.